CLINICAL TRIAL: NCT01604629
Title: Evaluation of Clinical Value of Standardized Protocol for Dose-reduction in Patients With Spondylarthropathies and Clinical Remission With Anti-TNF Therapy: Open-label, Controlled, Randomized, Multicenter Trial.
Brief Title: Evaluation of a Protocol for Dose Reduction in Patients With Spondylarthropathies and Clinical Remission With Anti-TNF
Acronym: REDES-TNF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Spanish Clinical Pharmacology Society (Other)
Collaborators: Spanish reumatology Society (Unknown)
Responsible Party: Principal Investigator, Dra. Caridad Pontes, Study coordinator, Spanish Clinical Pharmacology Society
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REDES-TNF/2012; 2011-005871-18 (EudraCT Number)
Record Dates: First submitted 2012-05-17; First posted 2012-05-24 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Spondylarthropathies
Keywords: Spondylarthropathies; Persistent clinical remission with anti-TNF therapy; Standardized protocol for dose reduction anti-TNF therapy
MeSH Terms: conditions — Spondylarthropathies | interventions — Adalimumab; Etanercept; golimumab; Infliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Reduced doses of anti-TNF (Experimental): Standardized schedule of reduced doses of anti-TNF, reached either through the interval spacing of administration (adalimumab, etanercept or golimumab) or reducing doses of infliximab
  Interventions: Drug: Reduced doses of anti-TNF
- Stable doses of anti-TNF (Active Comparator): Stable doses of anti-TNF according clinical practice based on approved summary product characteristics (SPC) and SER consensus about biological therapies in Ankylosing Spondylitis and other Spondylarthropathies, except Psoriatic Arthritis
  Interventions: Drug: Stable doses of anti-TNF

INTERVENTIONS:
Drug: Reduced doses of anti-TNF — Standardized schedule of reduced doses of anti-TNF, reached either through the interval spacing of administration (adalimumab, etanercept or golimumab) or reducing doses of infliximab
  Other Names: Adalimumab: 40 mg / 3 weeks; Etanercept: 50 mg / 10 days; Golimumab: 50 mg / 6 weeks; Infliximab: 3 mg/kg / 8 weeks
  Arms: Reduced doses of anti-TNF
Drug: Stable doses of anti-TNF — Stable doses of anti-TNF according clinical practice based on approved summary product characteristics (SPC) and SER consensus about biological therapies in Ankylosing Spondylitis and other Spondylarthropathies, except Psoriatic Arthritis
  Other Names: Adalimumab: 40 mg / 2 weeks; Etanercept: 25 mg / 3 days ó 50 mg /7 days; Golimumab: 50 mg / 4 weeks; Infliximab: 5 mg/kg / 6-8 weeks
  Arms: Stable doses of anti-TNF

SUMMARY:
The purpose of this study is to demonstrate that patients with Spondylarthropathies in remission under antiTNF therapy, can maintain the remission with a maintenance dose inferior to the currently recommended dose schedule.

DETAILED DESCRIPTION:
It has been shown that the withdrawal of treatment follows with a flare of the disease in a short time after the suspension but it has not been evaluated in controlled trials if remission could be maintained with a lower dose. A multicenter, national, open-label, randomized and controlled clinical trial of 3 years duration (2 years for inclusion + 1 year follow-up) is proposed to address this issue. The study will include 190 patients with Spondylarthropathies in stable treatment with any single anti-TNF agent and compliance with criteria of clinical remission for at least 4 months. Patients will be randomized to intervention or control arm, with stratification according to the antiTNF product thet were receiving prior to inclusion. Patients will be followed with the calendar of visits recommended by the Spanish Society of Rheumatology for clinical practice. The proposed hypothesis is of non-inferiority of the experimental arm with dose reduction versus the control arm with standard treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years
* Patients with Spondylarthropathies according ASAS group criteria.
* Patients under treatment with anti-TNF therapy (infliximab, adalimumab, etanercept, golimumab) who present established clinical remission
* Patients to give their informed consent to participate in the study

Exclusion Criteria:

* Patients with secondary Spondylarthropathies
* Patients with Spondylarthropathies and predominantly clinical of peripheral arthritis which receive anti-TNF therapy by peripheral symp tons.
* Patients with Spondylarthropathies and other associated diseases that hinders or modify the clinical evaluation of the patient (fibromyalgia, chronic inflammatory disorders…)
* Patients with bowel inflammatory disease
* Patients under chronic therapy with anti-TNF therapy who received the patterns of reduction that will be explored in the experimental group, or low doses or most spaced that those in the experimental group before study inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2012-07; Primary Completion 2015-04 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who are kept in the acceptable therapeutic objective according Spanish Rheumatology Society (SER) consensus, after one year | one year after inclusion
  Proportion of patients who are kept in the acceptable therapeutic objective according Spanish Society of Reumatology (SER) consensus (BASDAI < 4, global clinical impression by physician <4 and by patient < 4 and axial nocturnal pain <4) after one year

SECONDARY OUTCOMES:
Proportion of patients in remission one year after inclusion in the study | one year
  Proportion of patients in remission, defined as ASDAS-C score lower than than 1.3, after one year from inclusion in the study
Proportion of patients who experience a clinical reactivation | last study visit (up to 3 years or December 2014)
  Proportion of patients who experience a clinical reactivation, defined according criteria of active disease by Spanish Society of Reumatology (SER) consensus (BASDAI > 4, global clinical impression by physician >4 and at least one of three following criteria: patient impression >= 4, axial nocturnal pain (VAS) >= 4, and increased of acute phase reactants (reactive C protein (PCR) and/or erytrocyte sedimentation rate (ESR))
Proportion of patients who are kept in the acceptable therapeutic objective in the last study visit | last study visit (up to 3 years or December 2014)
  Proportion of patients who are kept in the acceptable therapeutic objective according Spanish Society of Reumatology (SER) consensus (BASDAI < 4, global clinical impression by physician <4 and by patient < 4 and axial nocturnal pain <4) in the last study visit
Proportion of patients who are kept in the ideal therapeutic objective in the last follow visit | last study visit (up to 3 years or December 2014)
  Proportion of patients who are kept in the ideal therapeutic objective according to the Spanish Society of Reumatology (SER) consensus (BASDAI < 2, global clinical impression by physician <2 and by patient < 2 ) in the last study visit
Time to clinical reactivation | last study visit (up to 3 years or December 2014)
  Time to clinical reactivation, defined according to the criteria of active disease by Spanish Society of Reumatology (SER) consensus, BASDAI + VAS and ASDAS, respectively
Withdrawal because of clinical requirement to modify the antiTNF treatment. | last study visit (up to 3 years or December 2014)
  Proportion of patients who are withdrawn from the study because of clinical requirement to modify the antiTNF treatment.
NSAIDs use | last study visit (up to 3 years or December 2014)
  NSAIDs use measured according semiquantitative Dougados criteria
Suspected Serious Adverse Reactions | last study visit (up to 3 years or December 2014)
  Proportion of patients who experience a Serious Adverse Event at least possibly related with anti-TNF therapy.
Time to Suspected Serious Adverse Reaction | last study visit (up to 3 years or December 2014)
  Time to Serious Adverse Events at least possibly related with anti-TNF therapy
Proportion of patients in remission after two years from inclusion in the study | 2 years
  Proportion of patients in remission, defined as ASDAS-C point less than 1.3, after two years from inclusion in the study

CONTACTS AND LOCATIONS:
Overall Officials: Gratacós Jordi, MD, PhD, Principal Investigator — Hospital de Sabadell - Corporació Sanitària i Universitaria Parc Taulí UAB
Locations (31):
- Spain (31):
  - Hospital Clínic Universitari Sant Joan d'Alacant, Alicante, Alacant
  - Hospital General de Llerena-Zafra, Llerena, Badajoz
  - Hospital Son Llàtzer, Palma de Mallorca, Balearic Islands
  - Hospital Clínic de Barcelona, Barcelona, Barcelona
  - Hospital Vall d'Hebron, Barcelona, Barcelona
  - IMIM-Hospital del Mar, Barcelona, Barcelona
  - Hospital Universitario de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Corporació Sanitària Parc Taulí, Sabadell, Barcelona
  - Hospital de Sant Joan Despí Moisès Broggi, Sant Joan Despí, Barcelona
  - Hospital Reina Sofía, Córdoba, Córdoba
  - Hospital Comarcal de Palamós, Palamós, Girona
  - Hospital Universitario de Guadalajara, Guadalajara, Guadalajara
  - Hospital Juan Canalejo, A Coruña, La Coruña
  - Hospital Universitario de Gran Canaria Dr. Negrín, Las Palmas de Gran Canaria, Las Palmas
  - Hospital Universitario Príncipe de Asturias, Alcalá de Henares, Madrid
  - Hospital Universitario Fundación Alcorcón, Alcorcón, Madrid
  - Hospital Clínico San Carlos, Madrid, Madrid
  - Hospital General Universitario Gregorio Marañón, Madrid, Madrid
  - Hospital Universitario 12 de Octubre, Madrid, Madrid
  - Hospital Universitario de La Princesa, Madrid, Madrid
  - Hospital Universitario La Paz, Madrid, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid, Madrid
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid
  - Hospital Universitario de Móstoles, Móstoles, Madrid
  - Hospital Universitario Virgen de la Arrixaca, Murcia, Murcia
  - Hospital Monte Naranco, Oviedo, Principality of Asturias
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Clínico de Salamanca, Salamanca, Salamanca
  - Hospital Universitario Virgen Macarena, Seville, Sevilla
  - Hospital Sant Pau i Santa Tecla, Tarragona, Tarragona
  - Hospital General de Valencia, Valencia, Valencia

REFERENCES:
- [Derived] Gratacos J, Pontes C, Juanola X, Sanz J, Torres F, Avendano C, Vallano A, Calvo G, de Miguel E, Sanmarti R; REDES-TNF investigators. Non-inferiority of dose reduction versus standard dosing of TNF-inhibitors in axial spondyloarthritis. Arthritis Res Ther. 2019 Jan 8;21(1):11. doi: 10.1186/s13075-018-1772-z. PMID 30621746